CLINICAL TRIAL: NCT07395453
Title: Assessments of Obsessive-compulsive Symptoms in Patients With Substances Use Disorder and Its Correlates
Brief Title: Assessments of Obsessive-compulsive Symptoms in Patients With Substances Use Disorder
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Refaat Sayed Ahmed, Resident of Neurology and Psychiatry, Assiut University
Other Study IDs: OCD in substances use disorder
Record Dates: First submitted 2025-12-04; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Obsessive - Compulsive Disorder; Obsessive Compulsive Disorder (OCD); Obsessive Compulsive Behavior; Substance Abuse Disorder; Substance Use
Keywords: obsessive-compulsive symptoms; substances use disorder
MeSH Terms: conditions — Compulsive Personality Disorder; Obsessive-Compulsive Disorder; Compulsive Behavior; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Substance Use Disorder Patients: Adults aged 18-50 years with a diagnosed substance use disorder (single or polysubstance) attending the inpatient or outpatient addiction management unit at Assiut University Hospital, assessed for obsessive-compulsive symptoms, psychiatric comorbidities, cognition, and quality of life using standardized scales and urine toxicology.
- Healthy Control Group: Adults aged 18-50 years without substance use disorder, recruited from relatives, friends, or hospital workers, matched on sociodemographic characteristics where feasible, and assessed with the same clinical and psychometric battery to compare obsessive-compulsive symptoms and related outcomes with the patient group.

SUMMARY:
This observational, cross-sectional case-control study evaluates obsessive-compulsive symptoms among adults with substance use disorder compared with a demographically similar control group without substance use disorder. Patients aged 18-50 years attending the addiction management inpatient and outpatient services at Assiut University Hospital, and healthy controls recruited from relatives, friends, and hospital staff, will complete structured clinical interviews, the Yale-Brown Obsessive-Compulsive Scale, and other standardized scales for psychiatric symptoms, cognition, and quality of life. The main objective is to estimate the prevalence and severity of obsessive-compulsive symptoms in substance use disorder and examine their associations with sociodemographic and clinical factors, addiction severity, and quality of life in the recovery stage.

DETAILED DESCRIPTION:
Substance use disorders and obsessive-compulsive disorder are chronic, relapsing conditions that share underlying neurobiological mechanisms related to compulsivity and have substantial impact on functioning and quality of life. Clinical experience and prior research suggest that obsessive-compulsive symptoms may be under-recognized among individuals with substance use disorders, where they can worsen psychiatric comorbidity, complicate treatment, and impair recovery.

The current study will recruit 102 adults aged 18-50 years, including 51 patients with a diagnosed substance use disorder (single or polysubstance) from the inpatient and outpatient addiction management unit at the Neuropsychiatry Department, Assiut University Hospital, and 51 control participants without substance use disorder drawn from relatives, friends, and hospital workers. All participants must be in a non-intoxicated, non-withdrawal state and able to provide informed consent; individuals with severe psychiatric disorders (such as schizophrenia, bipolar disorder, major depressive disorder with severe features, or anorexia nervosa), severe medical illness, or marked cognitive impairment will be excluded.

Data collection will include a structured sociodemographic and clinical sheet, brief psychiatric interview, and administration of validated instruments such as the Yale-Brown Obsessive-Compulsive Scale, Obsessive Compulsive Drug Use Scale, Symptom Checklist-90-R, Montreal Cognitive Assessment, and Hamilton scales for anxiety and depression, along with urine analysis for substances. The primary objective is to assess the correlation between obsessive-compulsive symptoms in patients with substance use disorder and both symptom severity and quality of life, while secondary objectives address compulsive aspects of addiction, craving in patients with obsessive-compulsive symptoms, and potential implications for management strategies.

ELIGIBILITY:
Inclusion Criteria:

--Adults aged 18-50 years.

* Willing and able to provide informed consent and participate in the study assessments.
* For the case group: patients with a diagnosed substance use disorder (single or polysubstance) attending the inpatient or outpatient addiction management unit at the Neuropsychiatry Department, Assiut University Hospital.
* For the control group: relatives, friends, or hospital workers without substance use disorder, recruited through invitation or advertisement.

Exclusion Criteria:

* Severe psychiatric comorbidities such as schizophrenia, major depressive disorder, bipolar disorder, or anorexia nervosa.
* Current intoxication or acute withdrawal state from substances.
* Severe medical conditions including end-stage renal disease, metastatic cancer, severe heart failure, or chronic obstructive pulmonary disease.
* Severe cognitive impairment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults aged 18-50 years attending the inpatient and outpatient addiction management unit at the Neuropsychiatry Department, Assiut University Hospital, with a diagnosed substance use disorder, and a comparison group of relatives, friends, or hospital workers without substance use disorder. Participants of both sexes who provide informed consent will be assessed once during the recovery (non-intoxication, non-withdrawal) stage using structured clinical interviews, standardized scales for obsessive-compulsive symptoms, psychiatric comorbidity, cognition, and global psychopathology, as well as urine toxicology.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Severity of Obsessive-Compulsive Symptoms in Patients with Substance Use Disorder Measured by Yale-Brown Obsessive Compulsive Scale (Y-BOCS) Total Score | Baseline (study enrollment during recovery stage defined as non-intoxication and non-withdrawal); single assessment
  Yale-Brown Obsessive Compulsive Scale (Y-BOCS) total score assessing severity of obsessive-compulsive symptoms in patients with substance use disorder. Scale ranges from 0 to 40 points, where higher scores indicate greater severity, assessed once at study enrollment during recovery stage defined as non-intoxication and non-withdrawal.